CLINICAL TRIAL: NCT01123382
Title: Electrical Stimulation for Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, John Chae, MD, Prof Vice Chair Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD059777 (NIH); R01HD059777 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Shoulder Pain
Keywords: Stroke; Shoulder pain; Electrical stimulation; Neuromuscular stimulation; Intramuscular stimulation
MeSH Terms: conditions — Stroke; Shoulder Pain | interventions — Home Infusion Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- IM Electrical Stimulation (IM ES) (Experimental): The IM ES Group will receive electrical stimulation treatment for three weeks (6 hrs daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period.
  Interventions: Device: Intramuscular Electrical Stimulator
- Usual Care (UC) (Active Comparator): The Usual Care Group will receive outpatient therapy for four weeks, coupled with prescribed daily home exercises.
  Interventions: Other: Outpatient Therapy

INTERVENTIONS:
Device: Intramuscular Electrical Stimulator — A sterile percutaneous IM electrode is implanted in the shoulder using a 20-gauge hypodermic needle and connected to an external cable. The exit site and electrode are covered by a bandage, but the cable extends out. After a one week stabilization period, the cable is connected to a stimulator. A self-adhesive surface electrode serves as the indifferent electrode. Stimulation intensity is set by the investigator. The prescription for daily stimulation treatment will be 6 hrs. The duty cycle and daily dose will remain constant throughout the treatment, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period will be 3 weeks, after which the electrode will be removed. Total time of electrode implantation is no more than 29 days.
  Arms: IM Electrical Stimulation (IM ES)
Other: Outpatient Therapy — Subjects will receive 8 hrs of outpatient therapy over a four week period from a treating therapist, coupled with prescribed daily home exercises. The therapist will implement an individualized treatment plan consistent with the needs of the participant.
  Arms: Usual Care (UC)

SUMMARY:
Post-stroke shoulder pain is a major rehabilitation problem affecting moderate to severely impaired stroke survivors. Surface electrical stimulation (ES) of muscles surrounding the hemiparetic shoulder has been demonstrated to be beneficial, but despite the evidence for therapeutic benefit, the clinical implementation of surface ES for poststroke shoulder pain has been difficult. In order to address the limitations of surface ES, the investigative team pioneered the development of percutaneous intramuscular (IM) ES for the treatment of post-stroke shoulder pain. However, prior to acceptance by the clinical community, additional gaps in the scientific and clinical knowledge need to be addressed. This study begins to do so. The primary objective is to estimate the relative pain reduction associated with IM ES vs. "usual care." We hypothesize that the IM ES group will exhibit a larger effect size with respect to pain reduction compared to "usual care". A secondary objective is to estimate the effect on health related QOL of IM ES vs. "usual care." Demonstration of improvement in QOL will validate the clinical relevance of the intervention. We hypothesize that the IM ES group will exhibit greater improvement in health related QOL compared to "usual care".

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain localized to the glenohumeral joint, subacromial area or deltoid insertion associated with any of the following conditions: a) rest; b) passive abduction or external rotation ROM; c) active abduction or external rotation ROM; or d) manual palpation
* weakness of shoulder abductors (≤4/5 on MRC if isolated movement is present)
* age ≥21-yrs
* time from stroke ≥ 3-mo
* shoulder pain onset after the most recent stroke
* duration of shoulder pain ≥ 3-mo
* severity of shoulder pain on BPI-SF 3 ≥4
* cognitive ability to fulfill study requirements [a) exhibit 3 object immediate and 30 minute recall; b) ability to use a numeric rating scale (using a 0-10 numeric rating scale) by correctly ranking the tightness they feel on the unaffected arm of 3 low-pressure inflations with a standard sphygmomanometer cuff which follow a predetermined sequence (20, 40 and 0 mm Hg); and c) ability to follow 3-stage commands]
* availability of a reliable adult who can check the skin and assist the participant with the treatment protocol
* willing and able to report severity of shoulder pain throughout the study period
* willing to make all scheduled study visits post-implantation.

Exclusion Criteria:

* evidence of joint or overlying skin infection
* insensate skin
* >1 opioid or nonopioid analgesics daily for shoulder pain
* daily intake of pain medications for any other chronic pain
* intra-articular or subacromial steroid injections to the shoulder in the previous 12-wks
* botulinum toxin injection to the trapezius, pectoralis or subscapularis muscle in the previous 12-wks
* receiving physical or occupational therapies for shoulder pain
* physician-diagnosed shoulder pathology symptomatic within the 5 yrs prior to CVA
* bleeding disorder
* INR>3.0 for those on warfarin [INR>3.0]
* poorly controlled diabetes [HbA1c>7.0]
* medical instability
* pregnancy
* uncontrolled seizures (>1/mo for 6-mo)
* uncompensated hemi-neglect
* severely impaired communication
* moderate to severe depression
* other confounding conditions such as ipsilateral upper limb lower motorneuron lesion, Parkinson's Disease, spinal cord injury, traumatic brain injury or multiple sclerosis
* other medical issues such as complex regional pain syndrome, bicipital tendonitis, myofacial pain syndrome, etc.
* the following cardiac conditions: a) history of arrhythmia with hemodynamic instability, such as ventricular tachycardia, supraventricular tachycardia and rapid ventricular response atrial fibrillation; b) any implantable stimulator such as demand pacemakers or defibrillators; and c) valvular heart disease including artificial valves (due to risk of infection and endocarditis)
* likely non-compliance factors such as distance from the center, inadequate social support, or psychiatric/psychologic factors

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chae, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu DT, Chae J, Walker ME, Fang ZP. Percutaneous intramuscular neuromuscular electric stimulation for the treatment of shoulder subluxation and pain in patients with chronic hemiplegia: a pilot study. Arch Phys Med Rehabil. 2001 Jan;82(1):20-5. doi: 10.1053/apmr.2001.18666. PMID 11239281
- [Background] Yu DT, Chae J, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Feldstein M, Fang ZP. Intramuscular neuromuscular electric stimulation for poststroke shoulder pain: a multicenter randomized clinical trial. Arch Phys Med Rehabil. 2004 May;85(5):695-704. doi: 10.1016/j.apmr.2003.07.015. PMID 15129391
- [Background] Chae J, Yu DT, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Fang ZP. Intramuscular electrical stimulation for hemiplegic shoulder pain: a 12-month follow-up of a multiple-center, randomized clinical trial. Am J Phys Med Rehabil. 2005 Nov;84(11):832-42. doi: 10.1097/01.phm.0000184154.01880.72. PMID 16244520
- [Background] Chae J, Ng A, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Intramuscular electrical stimulation for shoulder pain in hemiplegia: does time from stroke onset predict treatment success? Neurorehabil Neural Repair. 2007 Nov-Dec;21(6):561-7. doi: 10.1177/1545968306298412. Epub 2007 Mar 16. PMID 17369520
- [Derived] Wilson RD, Gunzler DD, Bennett ME, Chae J. Peripheral nerve stimulation compared with usual care for pain relief of hemiplegic shoulder pain: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Jan;93(1):17-28. doi: 10.1097/PHM.0000000000000011. PMID 24355994
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Groups:
- IM Electrical Stimulation (IM ES): The IM ES Group will receive electrical stimulation treatment for three weeks (6 hrs daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period.
  Intramuscular Electrical Stimulator: A sterile percutaneous IM electrode is implanted in the shoulder using a 20-gauge hypodermic needle and connected to an external cable. The exit site and electrode are covered by a bandage, but the cable extends out. After a one week stabilization period, the cable is connected to a stimulator. A self-adhesive surface electrode serves as the indifferent electrode. Stimulation intensity is set by the investigator. The prescription for daily stimulation treatment will be 6 hrs. The duty cycle and daily dose will remain constant throughout the treatment, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period will be 3 weeks, after which the electrode will be removed.
Period: Overall Study
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Started | 13 | 12
Received Intervention | 12 | 10
Completed | 11 | 6
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.0 [50.5 to 68.0] | 55.5 [50.0 to 62.5] | 55.0 [50.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 11
  African American | 7 | 6 | 13
  Hispanic/Latino | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 25
Shoulder pain > 18 mos [Count of Participants; unit: Participants] | 8 | 7 | 15
Time Since Stroke [Median (Inter-Quartile Range); unit: years] | 2.1 [0.9 to 4.0] | 2.3 [0.8 to 4.8] | 2.1 [0.9 to 4.6]

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Short Form
Description: The BPI is a pain questionnaire, which assesses both pain intensity (sensory dimension) and the interference (reactive dimension) of pain in daily activities. Pain intensity is measured on a 0 - 10 scale, with 0 being no pain and 10 being worst possible.
Time Frame: Baseline (Week 0); Start of Treatment (Week 1); End of Treatment (EOT, Week 4); EOT + 6 wks (Week 10); EOT + 12 wks (Week 16)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
units on a scale
  Week 0 | 7.5 (0.7) | 7.6 (0.7)
  Week 1 | 6.1 (0.7) | 6.8 (0.7)
  Week 4 | 2.6 (0.7) | 5.0 (0.8)
  Week 10 | 3.2 (0.7) | 6.1 (0.8)
  Week 16 | 3.0 (0.7) | 6.1 (0.8)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); To detect a minimum clinically important difference of 2 points2 on the BPI-SF3 with an anticipated standard deviation for each mean of 2.5, estimated from a prior study, with an alpha level of 0.05 and a power of 80%, for five waves of data, a sample size of 10 participants per group was necessary. With anticipated dropouts, a sample size of at least 12 participants per group was required; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — Group X time interaction; we included a random intercept for each individual participant. We used a first-order antedependent covariance structure

2. Secondary Outcome: ShoulderQ VGRS Scale
Description: The ShoulderQ Visual Graphics Rating Scale (VGRS) T is a structured questionnaire designed to assess severity of HSP at rest during the day, on movement, and at night on a 0-30 scale where higher numbers indicate greater pain.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
units on a scale
  Week 0 | 16.5 (1.7) | 16.5 (1.8)
  Week 1 | 14.8 (1.8) | 15.6 (1.8)
  Week 4 | 6.3 (1.8) | 11.0 (2.0)
  Week 10 | 6.7 (2.1) | 10.5 (2.2)
  Week 16 | 7.6 (2.4) | 13.1 (2.6)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — group x time interaction 0.059

3. Secondary Outcome: SF-36 Bodily Pain Component
Description: The SF-36v2 is a population-norm based health related quality of life measure, presented in T-scores where population average equals a score of 50 with a standard deviation of 10. Maximum is 100, with higher score indicating greater health realated quality of life.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
units on a scale
  Week 0 | 36.1 (1.9) | 36.4 (2.0)
  Week 1 | 41.2 (2.0) | 38.3 (2.1)
  Week 4 | 47.9 (2.2) | 44.9 (2.6)
  Week 10 | 48.3 (2.7) | 41.2 (3.1)
  Week 16 | 49.3 (3.3) | 46.9 (3.9)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.543, Mixed Models Analysis — group x time interaction 0.543

4. Secondary Outcome: Pain-free External ROM, Degrees
Description: Passive pain-free Externa ROM is a motor recovery measure. The subject was supine with the shoulder adducted with hand resting on the abdomen, elbow flexed, and with the humerus supported by the mat. The axis of a universal goniometer was centered on the olecranon process of the ulna projecting through the humeral shaft toward the humeral head. The subject's shoulder was externally rotated passively to the pain threshold, defined as the start of any pain. Pain at rest was recorded as 0 degrees.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
degrees
  Week 0 | 50.5 (14.4) | 26.7 (15.0)
  Week 1 | 56.2 (14.6) | 34.0 (15.2)
  Week 4 | 80.8 (14.6) | 43.7 (15.9)
  Week 10 | 77.0 (14.6) | 37.4 (15.6)
  Week 16 | 76.9 (14.6) | 41.5 (15.9)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.33, Mixed Models Analysis — group x time interaction 0.33

5. Secondary Outcome: Fugl-Myer Motor Assessment (FMA) - Upper Extremity
Description: The Fugl-Myer Motor Assessment (FMA) is a motor recovery measure. Volitional movement of the upper limb (shoulder, elbow, forearm, wrist, and hand) is examined in and out of synergies. Each item was graded on a 3-point ordinal scale and summed to provide a maximum score of 66, with higher scores indicating lower impairment.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
units on a scale
  Week 0 | 26.7 (6.6) | 23.0 (6.9)
  Week 1 | 27.2 (6.6) | 24.6 (6.9)
  Week 4 | 29.4 (6.6) | 24.1 (6.9)
  Week 10 | 29.6 (6.6) | 25.0 (6.9)
  Week 16 | 29.9 (6.6) | 26.2 (6.9)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.61, Mixed Models Analysis — group x time 0.61

6. Secondary Outcome: Pain Interference Questionnaire
Description: BPI-9 from Brief Pain Inventory, Short Form. Pain interference is on a 0 - 10 scale, with 0 being no interference, and 10 being complete interference.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
units on a scale
  Week 0 | 3.6 (0.7) | 5.0 (0.7)
  Week 1 | 2.3 (0.7) | 4.6 (0.7)
  Week 4 | 0.8 (0.7) | 2.1 (0.8)
  Week 10 | 0.8 (0.7) | 3.0 (0.8)
  Week 16 | 1.1 (0.7) | 3.5 (0.8)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.398, Mixed Models Analysis — group x time interaction 0.398

7. Secondary Outcome: Isometric Shoulder Abduction Moment, Ratio Affected to Unaffected
Description: A measure of isometric strength in response to audio cue. Isometric shoulder abduction moment was measured with a Biodex Biomechanical Measurement System (Biodex Medical Systems, Shirley, NY). The average moment during the last second of the audible tone was calculated for each trial and those values were averaged over the three trials. Subjects underwent testing of both shoulders, non-paretic side first, and the results are presented as the ratio of the paretic shoulder to the non-paretic shoulder to decrease the influence of intra-subject variability between measurements.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio of affected to unaffected arm
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
ratio of affected to unaffected arm
  Week 0 | 0.3 (0.1) | 0.3 (0.1)
  Week 1 | 0.4 (0.1) | 0.3 (0.1)
  Week 4 | 0.4 (0.1) | 0.3 (0.1)
  Week 10 | 0.5 (0.1) | 0.3 (0.1)
  Week 16 | 0.5 (0.1) | 0.4 (0.1)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.46, Mixed Models Analysis — group x time interaction 0.46

8. Secondary Outcome: Delay in Initiation of Shoulder Abduction EMG Activity
Description: Electromyographic activity from the deltoid was also measured during the isometric abduction moment trials. Surface EMG recording electrodes (2 cm x 2 cm) were placed over the deltoid muscle and spaced approximately 4 cm apart. The EMG amplifier gain was adjusted to record as high-fidelity an EMG signal as possible during shoulder abduction. Delay of initiation (DOI) was defined as the duration between onset of the audibe tone and the onset of EMG signal. Raw EMG signals were analyzed visually to determine the earliest rise in EMG activity relative to steady state for delay of initiation. The mean DOI of the three trials were calculated, and the ratio of the paretic to non-paretic shoulder DOI were used as summary metrics.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio of affected to unaffected arm
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
ratio of affected to unaffected arm
  Week 0 | 1.4 (0.2) | 1.6 (0.2)
  Week 1 | 1.3 (0.2) | 1.3 (0.3)
  Week 4 | 1.2 (0.2) | 1.4 (0.3)
  Week 10 | 1.2 (0.2) | 1.2 (0.3)
  Week 16 | 1.4 (0.2) | 1.2 (0.3)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.59, Mixed Models Analysis — group x time interaction 0.59

9. Secondary Outcome: Delay in Termination of Shoulder Abduction EMG Activity
Description: Electromyographic activity from the deltoid was also measured during the isometric abduction moment trials. Surface EMG recording electrodes (2 cm x 2 cm) were placed over the deltoid muscle and spaced approximately 4 cm apart. The EMG amplifier gain was adjusted to record as high-fidelity an EMG signal as possible during shoulder abduction. Delay of termination (DOT) was defined as the duration between cessation of the audible tone and return of the EMG signal to baseline. Raw EMG signals were analyzed visually to determine the earliest rise in EMG activity relative to steady state for delay of initiation, and return to steady for delay of termination. The mean DOT of the three trials were calculated, and the ratio of the paretic to non-paretic shoulder DOT were used as summary metrics.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio of affected to unaffected arm
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Number analyzed (Participants) | 13 | 12
ratio of affected to unaffected arm
  Week 0 | 2.3 (0.5) | 1.3 (0.6)
  Week 1 | 2.6 (0.6) | 3.7 (0.6)
  Week 4 | 1.7 (0.6) | 2.0 (0.7)
  Week 10 | 1.9 (0.7) | 1.5 (0.5)
  Week 16 | 1.7 (0.5) | 2.6 (0.7)
Statistical Analysis 1: Comparison: IM Electrical Stimulation (IM ES) vs Usual Care (UC); Test type: Superiority or Other; p = 0.69, Mixed Models Analysis — group x time interaction 0.69

ADVERSE EVENTS:
Arm/Group | IM Electrical Stimulation (IM ES) | Usual Care (UC)
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/12
Other Adverse Events (participants affected / at risk) | 10/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM Electrical Stimulation (IM ES) (N=13) | Usual Care (UC) (N=12)
Chest pain, hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Headache, hospitalization (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IM Electrical Stimulation (IM ES) (N=13) | Usual Care (UC) (N=12)
Electrode dislodgement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/0
Retained Electrode Fragment (Musculoskeletal and connective tissue disorders) | 3 (3) | 0/0
Pruritus at electrode or bandage site (Musculoskeletal and connective tissue disorders) | 6 (6) | 0/0
Pain after electrode implantation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No